CLINICAL TRIAL: NCT04605588
Title: A Triple Combination Antiviral Coronavirus Therapy (TriACT) RCT Comparing Nitazoxanide, Ribavirin and Hydroxychloroquine vs. Placebo
Brief Title: A Triple Combination Antiviral Coronavirus Therapy (TriACT) for COVID-19
Acronym: TriACT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of participants willing to enroll
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: SynaVir (Industry)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Distinguished Professor of Medicine, Robert Wood Johnson Medical School, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2020001862
Record Dates: First submitted 2020-10-26; First posted 2020-10-28 (Actual); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV Infection; Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — nitazoxanide; Ribavirin; Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study medication will be tablets/capsules containing either active drug or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Study Drug (Active Comparator): 5 day dosing of Nitazoxanide, Ribavirin & Hydroxychloroquine sulfate
  Interventions: Drug: Nitazoxanide; Drug: Ribavirin; Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): 5 day dosing of placebo
  Interventions: Drug: Placebo Nitazoxanide; Drug: Placebo Ribavirin; Drug: Placebo Hydroxychloroquine

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide (500 mg po BID for day 1and then 500 mg BID for 4 days)
  Arms: Active Study Drug
Drug: Placebo Nitazoxanide — Placebo Nitazoxanide (500 mg po BID for day 1and then 500 mg BID for 4 days)
  Arms: Placebo
Drug: Ribavirin — Ribavirin (600 mg po BID for day 1and then 400 mg BID for 4 days)
  Arms: Active Study Drug
Drug: Placebo Ribavirin — Placebo Ribavirin (600 mg po BID for day 1and then 400 mg BID for 4 days)
  Arms: Placebo
Drug: Hydroxychloroquine — Hydroxychloroquine sulfate (400 mg po BID for day 1 and then 200 mg BID for 4 days)
  Arms: Active Study Drug
Drug: Placebo Hydroxychloroquine — Placebo Hydroxychloroquine sulfate (400 mg po BID for day 1 and then 200 mg BID for 4 days)
  Arms: Placebo

SUMMARY:
New outpatient treatments for COVID-19 are urgently needed. There is some evidence that a combination of three medications currently used to treat other viral infections could be effective in fighting this new virus. The purpose of this trial is to evaluate the efficacy of Nitazoxanide (NTZ), Ribavirin (RBV) and Hydroxychloroquine (HCQ) versus placebo in participants with proven SARS-CoV-2 infection

The study will enroll 70 participants within the 7 days after having been diagnosed with coronavirus infection. The purpose is to determine if those randomized to 5-day dosing with the three medication combination have decreased viral load and severity of illness in the 10 days following treatment as compared to those taking placebo. Participants will be actively followed for 28 days.

DETAILED DESCRIPTION:
Participants will be randomized into one of two treatment plans

* Triple combination:

  * Nitazoxanide (500 mg po BID for day 1and then 500 mg BID for 4 days)
  * Ribavirin (600 mg po BID for day 1and then 400 mg BID for 4 days)
  * Hydroxychloroquine sulfate (400 mg po BID for day 1 and then 200 mg BID for 4 days)
* No active Medication:

  * Placebo administered according to the above schedule

Viral load (qPCR via nasal swab) will be assessed at baseline (day 0) as well as at days 3, 6, and 10 to monitor response to antiviral treatment. Immune status will be determined by antibody testing of blood collected at baseline and day 28. Symptom questionnaires will be completed daily for 10 days and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Documented SARS-CoV-2 infection by qPCR assay performed within the past 7 days

Exclusion Criteria:

* COVID-19 symptoms requiring hospitalization
* PO2 < 92%
* Short of breath at time of enrollment
* Retinal eye disease
* Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency
* Known chronic kidney disease, stage - 5 or receiving dialysis
* Current use of:

  * Class 3 AAD (amiodarone, dronaderone, dofetilide, sotalol)
  * Class 1A AAD (procainamide, quinidine, disopyramide)
  * Flecainide
  * SSRI: citalopram (Celexa), Escitalopram (Lexapro)
  * chlorpromazine
  * Cilostazol (Pletal)
  * Donepezil (Aricept)
  * Droperidol
  * Fluoconazole
  * Methadone
  * Ondansetron (Zofran)
  * Thioridazine
  * Macrolides (clarithromycin, erythromycin)
  * Fluroquinolones (ciprofloxacin, levofloxacin, moxifloxacin)
  * Tamoxifen
* Pregnancy or women who are breast feeding
* Inability to tolerate oral medications
* Allergy or prior adverse reaction to either hydroxychloroquine sulfate, ribavirin, or nitazoxanide
* Allergy to adhesives
* QTc interval > 450 mSEC for men and women
* History of Torsade de Pointes VT or prior cardiac arrest or congenital long QT interval
* Non-English-speaking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Study Drug | Placebo
Started | 2 | 5
Completed | 1 | 5
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Study Drug | Placebo | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (2.8) | 44 (15.0) | 42 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Decline in Viral Load Over the 10 Days After Randomization
Description: qPCR measured via nasal swab
Time Frame: 10 days after randomization
Population: This trial was terminated due to lack of enrollment. A total of 7 participants were randomized. Study outcome was to be response to antiviral treatment (rate of decline in viral load over the 10 days after randomization) as measured via nasal swab qPCR analysis. Based on the lack of enrollment, the swab analysis was not performed.
Arm/Group | Active Study Drug | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | Active Study Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04605588/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT04605588/ICF_000.pdf